CLINICAL TRIAL: NCT06574490
Title: Effectiveness of Myofunctional Therapy in Children With Open Bite - a Randomized Clinical Trial
Brief Title: Myofunctional Therapy in Open Bite - RCT
Acronym: Myofunctional
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Piotr Fudalej (Other)
Responsible Party: Sponsor-Investigator, Piotr Fudalej, Professor, Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1072.6120.39.2024
Record Dates: First submitted 2024-08-13; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Open Bite
Keywords: open bite; child; myofunctional; myotherapy; exercises
MeSH Terms: conditions — Open Bite; Motor Activity | interventions — Myofunctional Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofunctional + (Experimental): A series of myofunctional exercises
  Interventions: Procedure: Myofunctional therapy (+)
- Myofunctional - (Active Comparator): No exercises
  Interventions: Procedure: Myofunctional therapy (-)

INTERVENTIONS:
Procedure: Myofunctional therapy (+) — A series of myofunctional exercises performed in 10-20 sessions over 6 months
  Arms: Myofunctional +
Procedure: Myofunctional therapy (-) — NO exercises; A series of myofunctional exercises performed in 10-20 sessions over 6 months is delayed by 1 year
  Arms: Myofunctional -

SUMMARY:
The goal of this clinical trial is to learn if myofunctional therapy in 6-10-year-old children with infant type of swallowing and open bite is effective.

Primary hypothesis: myofunctional therapy results in correction of open bite Researchers will compare a group in which myofunctional therapy is performed for 6 months to a group in which myoufunctional therapy will be delayed by 1 year.

Participants will exercise according to a pre-established regimen and schedule

ELIGIBILITY:
Inclusion Criteria:

* generally healthy children aged 6-10 years,
* infant swallowing type,
* open anterior occlusion (i.e. no contact between the maxillary and mandibular medial incisors),
* mixed dentition

Exclusion Criteria:

* finger sucking habit (or similar) occurring within the last 6 months,
* previous myofunctional therapy,
* upper airway obstruction,
* congenital craniofacial developmental disorder,
* connective tissue or muscle disease,
* macroglossia,
* ankyloglossia,
* mental retardation

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Overbite | 12months
  presence positive vertical (i.e. the upper teeth overlap the lower teeth) and horizontal (i.e. the upper teeth are positioned in front of the lower teeth) occlusion

SECONDARY OUTCOMES:
Swallowing pattern | 12 months
  swallowing pattern (infant, adult or mixed)
Articulation | 12 months
  articulation of l,n,d,t,s sounds.